CLINICAL TRIAL: NCT03407144
Title: An Open-label, Uncontrolled, Multicenter Phase II Trial of MK-3475 (Pembrolizumab) in Children and Young Adults With Newly Diagnosed Classical Hodgkin Lymphoma With Inadequate (Slow Early) Response to Frontline Chemotherapy (KEYNOTE 667)
Brief Title: Safety and Efficacy of Pembrolizumab (MK-3475) in Children and Young Adults With Classical Hodgkin Lymphoma (MK-3475-667/KEYNOTE-667)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-667; MK-3475-667 (Other: MSD Protocol Number); 2023-504821-38 (Registry Identifier: EU CT); 2017-001123-53 (EudraCT Number)
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Hodgkin Lymphoma
Keywords: Programmed Death-1 (PD-1); PD1; Programmed Death-Ligand 1 (PD-L1); PDL1
MeSH Terms: conditions — Hodgkin Disease | interventions — pembrolizumab; Doxorubicin; Vinblastine; Dacarbazine; Cyclophosphamide; Vincristine; Prednisone; Prednisolone; Bleomycin; Etoposide; etoposide phosphate; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + AVD (Group 1) (Experimental): After receiving two 4-week cycles of ABVD (doxorubicin, bleomycin, vinblastine and dacarbazine) induction therapy, SER participants in Group 1 will receive pembrolizumab 2 mg/kg up to a maximum of 200 mg (3 to 17 years of age) or 200 mg (18 to 25 years of age) on Day 1 of each 3-week cycle (Q3W) in combination with two cycles of AVD chemotherapy (doxorubicin 25 mg/m^2, vinblastine 6 mg/m^2 and dacarbazine 375 mg/m^2 on Days 1 and 15; cycle frequency every 4 weeks [Q4W]). All SERs in Group 1 will receive radiotherapy (RT) after completing AVD chemotherapy.
  Interventions: Biological: pembrolizumab; Drug: doxorubicin; Drug: vinblastine; Drug: dacarbazine; Drug: bleomycin; Radiation: Radiotherapy (RT)
- Pembrolizumab + COPDAC-28 (Group 2) (Experimental): After receiving two 4-week cycles of OEPA (vincristine, etoposide/etopophos, prednisone/prednisolone and doxorubicin) induction therapy, SER participants in Group 2 will receive pembrolizumab 2 mg/kg up to a maximum of 200 mg (3 to 17 years of age) or 200 mg (18 to 25 years of age) Q3W, in combination with 4 cycles of COPDAC-28 chemotherapy (cyclophosphamide 500 mg/m^2 on Days 1 and 8, vincristine 1.5 mg/m^2 with maximum single dose 2 mg on Days 1 and 8, prednisone/prednisolone 40 mg/m^2/day divided in 3 doses on Days 1 to 15, dacarbazine 250 mg/m^2 on Days 1 to 3; cycle frequency Q4W). SERs in Group 2 will receive RT if they have a positive Positron Emission Tomography (PET) response after completing COPDAC-28 chemotherapy.
  Interventions: Biological: pembrolizumab; Drug: doxorubicin; Drug: dacarbazine; Drug: cyclophosphamide; Drug: vincristine; Drug: prednisone/prednisolone; Drug: etoposide; Radiation: Radiotherapy (RT)

INTERVENTIONS:
Biological: pembrolizumab — 2 mg/kg intravenous (IV) up to a max of 200 mg (3 to 17 years of age) or 200 mg IV (18 to 25 years of age); cycle frequency Q3W
  Other Names: MK-3475
Drug: doxorubicin — 25 mg/m^2 IV on Days 1 and 15 as part of ABVD induction therapy (cycle frequency: Q4W, Group 1)
  40 mg/m^2 IV on Days 1 and 15 as part of OEPA induction therapy (cycle frequency: Q4W, Group 2)
  25 mg/m^2 IV on Days 1 and 15 as part of AVD chemotherapy (cycle frequency: Q4W, Group 1)
Drug: vinblastine — 6 mg/m^2 IV on Days 1 and 15 as part of ABVD induction therapy (cycle frequency: Q4W, Group 1)
  6 mg/m^2 IV on Days 1 and 15 as part of AVD chemotherapy (cycle frequency: Q4W, Group 1)
  Arms: Pembrolizumab + AVD (Group 1)
Drug: dacarbazine — 375 mg/m^2 IV on Days 1 and 15 as part of ABVD induction therapy (cycle frequency: Q4W, Group 1)
  375 mg/m^2 IV on Days 1 and 15 as part of AVD chemotherapy (cycle frequency: Q4W, Group 1)
  250 mg/m^2 IV on Days 1 to 3 as part of COPDAC-28 chemotherapy (cycle frequency: Q4W, Group 2)
Drug: cyclophosphamide — 500 mg/m^2 IV on days 1 and 8 as part of COPDAC-28 chemotherapy (cycle frequency: Q4W, Group 2)
  Arms: Pembrolizumab + COPDAC-28 (Group 2)
Drug: vincristine — 1.5 mg/m^2 IV with maximum single dose 2 mg on Days 1, 8, and 15 as part of OEPA induction therapy (cycle frequency: Q4W, Group 2)
  1.5 mg/m^2 IV with maximum single dose 2 mg on Days 1 and 8 as part of COPDAC-28 chemotherapy (cycle frequency: Q4W, Group 2)
  Arms: Pembrolizumab + COPDAC-28 (Group 2)
Drug: prednisone/prednisolone — 60 mg/m^2/day orally divided in 3 doses on Days 1 to 15 as part of OEPA induction therapy (cycle frequency: Q4W, Group 2)
  40 mg/m^2/day orally divided in 3 doses on Days 1 to 15 as part of COPDAC-28 chemotherapy (cycle frequency: Q4W, Group 2)
  Arms: Pembrolizumab + COPDAC-28 (Group 2)
Drug: bleomycin — 10 units/m^2 IV on Days 1 and 15 as part of ABVD induction therapy (cycle frequency: Q4W, Group 1)
  Arms: Pembrolizumab + AVD (Group 1)
Drug: etoposide — 125 mg/m^2 IV on Days 1 to 5 as part of OEPA induction therapy (cycle frequency: Q4W, Group 2)
  Other Names: Etoposide Phosphate
  Arms: Pembrolizumab + COPDAC-28 (Group 2)
Radiation: Radiotherapy (RT) — RT administered daily, dose dependent on randomization group and disease response.

SUMMARY:
This study will examine the safety and efficacy of pembrolizumab (MK-3475) in combination with chemotherapy in children and young adults with newly diagnosed classical Hodgkin Lymphoma (cHL) who are slow early responders (SERs) to frontline chemotherapy.

DETAILED DESCRIPTION:
Group 1 will consist of low-risk participants with cHL Stages IA, IB and IIA without bulky disease. Group 2 will consist of high-risk participants with cHL Stages IIEB, IIIEA, IIIEB, IIIB, IVA and IVB.

ELIGIBILITY:
Inclusion Criteria:

* Group 1: Must have newly diagnosed, pathologically confirmed classical Hodgkin Lymphoma (cHL) at Stages IA, IB and IIA without bulky disease. Group 2: Must have newly diagnosed, pathologically confirmed cHL at Stages IIEB, IIIEA,IIIEB, IIIB, IVA and IVB
* Has measurable disease per investigator assessment.
* Male participants are eligible to participate if they agree to the following during the intervention period: refrain from donating sperm plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent or must agree to use contraception per protocol unless confirmed to be azoospermic.
* Female participants who are not pregnant or breastfeeding, and who are either not a woman of childbearing potential (WOCBP), or are a WOCBP who agrees to use approved contraception during the intervention period and for at least 120 days after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period.
* Performance status: Lansky Play-Performance Scale ≥50 for children up to 16 years of age OR Karnofsky score ≥50 for participants ≥ 16 years of age
* Has adequate organ function

Exclusion Criteria:

* Has undergone solid organ transplant at any time, or prior allogeneic hematopoietic stem cell transplantation within the last 5 years
* WOCBP who has a positive urine pregnancy test within 24 hours before the first dose of study treatment
* Baseline left ventricular ejection fraction value <50% or shortening fraction of <27%
* Has received prior therapy with an anti-Programmed Death (PD)-1, anti-Programmed Death-Ligand 1 (PD-L1), or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor or has previously participated in a MSD pembrolizumab (MK-3475) clinical study
* Has received any prior systemic anti-cancer therapy,including investigational agents for current diagnosis before randomization
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration
* Has a diagnosis of lymphocyte-predominant Hodgkin Lymphoma (HL)
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab
* Has a known additional malignancy that is progressing or requires active treatment within the past 3 years
* Has radiographically detectable central nervous system metastases and/or carcinomatous meningitis as assessed by local site investigator at the time of diagnosis
* Has severe hypersensitivity (≥Grade 3) to any study therapies including any excipients
* An active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study
* Participants who have not adequately recovered from major surgery or have ongoing surgical complications

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 340 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2027-02-13 (Estimated); Study Completion 2027-02-13 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in SER Participants By Risk Group (Low, High) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 8 years
  ORR is defined as the percentage of SER participants who have a Complete Response ([CR], disappearance of all evidence of disease) or Partial Response ([PR], regression of measurable disease and no new sites) using IWG revised response criteria and determined by BICR. The ORR will be estimated by risk group in SER participants.

SECONDARY OUTCOMES:
Rate of Positron Emission Tomography (PET) Scan Negativity in SER Participants By Risk Group (Low, High) After AVD or COPDAC-28 Chemotherapy | Up to approximately 8 years
  The rate of PET negativity for SER participants is the percentage of participants with PET negativity (defined as Deauville score 1, 2 or 3) after two cycles of AVD (Group 1) or four cycles of COPDAC-28 (Group 2), in combination with pembrolizumab. The Deauville 5-point scoring system is an internationally accepted and utilized five-point scoring system for the Fluorodeoxyglucose (FDG) avidity of a Hodgkin's lymphoma or Non-Hodgkin's lymphoma tumor mass as seen on FDG PET scan: Score 1= No uptake above the background, Score 2= Uptake ≤ mediastinum, Score 3= Uptake > mediastinum but ≤ liver, Score 4= Uptake moderately increased compared to the liver at any site, Score 5= Uptake markedly increased compared to the liver at any site or new lesions, Score X= New areas of uptake unlikely to be related to lymphoma. In the present study, scores of 1, 2 and 3 are considered to be negative and scores of 4 and 5 are considered to be positive.
Event-Free Survival (EFS) in SER Participants By Risk Group (Low, High) as Assessed by BICR | Up to approximately 8 years
  EFS is defined as the time from study enrollment to the first documented disease progression or recurrence, or death due to any cause, whichever occurs first. Progression/disease recurrence will be determined by BICR using IWG criteria.
Overall Survival (OS) in SER Participants By Risk Group (Low, High) | Up to approximately 8 years
  OS is defined as the time from study enrollment to death due to any cause. Participants without documented death will be censored at the date of the last follow-up.
Exposure to Radiotherapy (RT) in SER Participants By Risk Group (Low, High) | Up to approximately 8 years
  The frequency of RT received by eligible participants (positive PET response, i.e. Deauville score of 4 or 5) will be reported.
Rate of PET Scan Negativity In Group 1 Participants After ABVD Induction Therapy | Up to approximately 8 years
  The rate of PET negativity for Group 1 participants is the percentage of participants with PET negativity (defined as Deauville score 1, 2 or 3) after two cycles of ABVD induction as per investigator assessment. The Deauville 5-point scoring system is an internationally accepted and utilized five-point scoring system for the FDG avidity of a Hodgkin's lymphoma or Non-Hodgkin's lymphoma tumor mass as seen on FDG PET scan: Score 1= No uptake above the background, Score 2= Uptake ≤ mediastinum, Score 3= Uptake > mediastinum but ≤ liver, Score 4= Uptake moderately increased compared to the liver at any site, Score 5= Uptake markedly increased compared to the liver at any site or new lesions, Score X= New areas of uptake unlikely to be related to lymphoma. In the present study, scores of 1, 2 and 3 are considered to be negative and scores of 4 and 5 are considered to be positive.
EFS in Rapid Early Responder (RER) Participants By Risk Group (Low, High) as Assessed by Investigator | Up to approximately 8 years
  EFS is defined as the time from study enrollment to the first documented disease progression or recurrence, or death due to any cause, whichever occurs first. Progression/disease recurrence will be determined by the investigator.
OS in RER Participants By Risk Group (Low, High) | Up to approximately 8 years
  OS is defined as the time from study enrollment to death due to any cause. Participants without documented death will be censored at the date of the last follow-up.
Serum Thymus and Activation-Regulated Chemokine (TARC) Levels in SER Participants By Risk Group (Low, High) | Up to approximately 8 years
  Serum TARC levels will be measured and evaluated as a potential biomarker in SER participants by risk group at screening, early, and late response assessments.
Number of SER Participants Experiencing an Adverse Event (AE) By Risk Group (Low, High) | Up to approximately 8 years
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of SER participants who experience an AE will be reported for each arm.
Number of SER Participants Discontinuing Study Treatment Due to AEs By Risk Group (Low, High) | Up to approximately 8 years
  An AE is any untoward medical occurrence in a participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment. The number of SER participants who discontinue study treatment due to an AE will be reported for each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (93):
- United States (47):
  - Children's Hospital of Alabama ( Site 0023), Birmingham, Alabama
  - Phoenix Childrens Hospital ( Site 0034), Phoenix, Arizona
  - Arkansas Children's Hospital ( Site 0046), Little Rock, Arkansas
  - Kaiser - Orange County ( Site 0084), Anaheim, California
  - Kaiser Permanente ( Site 0082), Downey, California
  - Kaiser - Fontana ( Site 0083), Fontana, California
  - MemorialCare Health System - Long Beach Medical Center-Cherese Mari Laulhere Children's Village ( Si, Long Beach, California
  - Kaiser Permanente Downey Medical Center ( Site 0024), Los Angeles, California
  - Kaiser Permanente - Oakland ( Site 0047), Oakland, California
  - Kaiser Permanente - Roseville ( Site 0080), Roseville, California
  - Kaiser Permanente - Santa Clara ( Site 0079), Santa Clara, California
  - Children's Hospital - Colorado ( Site 0028), Aurora, Colorado
  - Connecticut Children's Medical Center ( Site 0045), Hartford, Connecticut
  - Yale Cancer Center ( Site 0061), New Haven, Connecticut
  - Children's National Medical Center ( Site 0090), Washington D.C., District of Columbia
  - University of Florida ( Site 0051), Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital ( Site 0048), Hollywood, Florida
  - Arnold Palmer Hospital ( Site 0065), Orlando, Florida
  - Children's Healthcare of Atlanta at Egleston ( Site 0033), Atlanta, Georgia
  - University of Chicago ( Site 0066), Chicago, Illinois
  - Riley Hospital for Children ( Site 0091), Indianapolis, Indiana
  - University of Kentucky Markey Cancer Center ( Site 0057), Lexington, Kentucky
  - University of Louisville-Norton Children's Hospital ( Site 0059), Louisville, Kentucky
  - Johns Hopkins University ( Site 0025), Baltimore, Maryland
  - Children's Hospital of Michigan ( Site 0056), Detroit, Michigan
  - Karmanos Cancer Institute ( Site 0002), Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota ( Site 0036), Minneapolis, Minnesota
  - St. Louis Children's Hospital ( Site 0038), St Louis, Missouri
  - Alliance for Childhood Diseases ( Site 0064), Las Vegas, Nevada
  - Hackensack University Medical Center ( Site 0026), Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey ( Site 0027), New Brunswick, New Jersey
  - Roswell Park Cancer Institute ( Site 0040), Buffalo, New York
  - Cohen Children's Medical Center of New York ( Site 0052), New Hyde Park, New York
  - Columbia University/Herbert Irving Cancer Center ( Site 0063), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0060), New York, New York
  - Weill Cornell Medicine ( Site 0032), New York, New York
  - UNC Lineberger Comprehensive Cancer ( Site 0044), Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center ( Site 0035), Cincinnati, Ohio
  - Nationwide Children's Hospital ( Site 0037), Columbus, Ohio
  - St. Francis Hospital Cancer Center ( Site 0001), Greenville, South Carolina
  - Vanderbilt University Medical Center-Ingram Cancer Center ( Site 0054), Nashville, Tennessee
  - Dell Children's Medical Center Of Central Texas ( Site 0058), Austin, Texas
  - Children's Medical Center ( Site 0030), Dallas, Texas
  - Texas Children's Hospital ( Site 0042), Houston, Texas
  - Methodist HealthCare System of San Antonio Clinical Trials Office, Texas Transplant Institute ( Site, San Antonio, Texas
  - Inova Fairfax Hospital ( Site 0031), Falls Church, Virginia
  - Seattle Childrens Hospital ( Site 0022), Seattle, Washington
- Brazil (3):
  - Hospital Erasto Gaertner-CEPEP - Pesquisa Clínica ( Site 0507), Curitiba, Paraná
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 0510), Natal, Rio Grande do Norte
  - Instituto de Oncologia Pediatrica - GRAACC - Unifesp ( Site 0500), São Paulo
- Colombia (4):
  - Hospital Pablo Tobon Uribe-Hematology ( Site 0565), Medellín, Antioquia
  - Organizacion Clinica Bonnadona-Prevenir S.A.S. ( Site 0529), Barranquilla, Atlántico
  - Instituto Nacional De Cancerologia ( Site 0566), Bogotá, Bogota D.C.
  - Oncomédica S.A.S ( Site 0527), Montería, Departamento de Córdoba
- Fakultni nemocnice v Motole ( Site 0356), Prague, Czechia
- France (7):
  - Institut d'Hematologie-Oncologie Pediatrique (IHOP) ( Site 0448), Lyon, Auvergne-Rhône-Alpes
  - CHU de Marseille Hopital de la Timone Enfants ( Site 0449), Marseille, Bouches-du-Rhone
  - CHU de Bordeaux. Hopital Pellegrin ( Site 0447), Bordeaux, Gironde
  - Hôpital Jeanne de Flandre ( Site 0450), Lille, Nord
  - Institut Gustave Roussy ( Site 0445), Villejuif, Val-de-Marne
  - Hopital d'Enfants Armand Trousseau ( Site 0443), Paris
  - Hopital Universitaire Robert Debre ( Site 0446), Paris
- Germany (5):
  - Klinikum der Universitaet Muenchen-Campus Innenstadt ( Site 0414), Munich, Bavaria
  - Universitaetsklinikum Giessen und Marburg GmbH ( Site 0411), Giessen, Hesse
  - Universitaetsklinikum Essen ( Site 0415), Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus-Pädiatrische Hämatologie und Onkologie ( Sit, Münster, North Rhine-Westphalia
  - Charite-Universitaetsmedizin Berlin Campus Virchow-Klinikum ( Site 0413), Berlin
- Greece (3):
  - Athens Childrens Hospital Aglaia Kyriakou ( Site 0361), Athens, Attica
  - University of Athens - Aghia Sophia Childrens Hospital ( Site 0362), Athens, Attica
  - University General Hospital of Thessaloniki "AHEPA" ( Site 0363), Thessaloniki, Central Macedonia
- Guatemala (3):
  - Oncomedica ( Site 0545), Guatemala City
  - Unidad Nacional de Oncologia Pediatrica ( Site 0542), Guatemala City
  - Medi-K Cayala ( Site 0544), Guatemala City
- Italy (5):
  - Universita degli Studi di Roma La Sapienza ( Site 0403), Roma, Abruzzo
  - Centro di Riferimento Oncologico CRO ( Site 0404), Aviano, Pordenone
  - Azienda Ospedaliera Santobono - Pausilipon ( Site 0402), Napoli
  - IRCCS Ospedale Pediatrico Bambino Gesu ( Site 0400), Roma
  - Ospedale Infantile Regina Margherita ( Site 0401), Torino
- Mexico (4):
  - Hospital Infantil de Mexico Federico Gomez ( Site 0535), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" ( Site 0531), Monterrey, Nuevo León
  - UMAE Hospital de Especialidades - CMN La Raza ( Site 0536), Azcapotzalco
  - Hematologica Alta Especialidad ( Site 0532), Huixquilucan
- Prinses Maxima Centrum ( Site 0461), Utrecht, Netherlands
- Narodny ustav detskych chorob ( Site 0372), Bratislava, Bratislava Region, Slovakia
- South Africa (3):
  - Wits Clinical Research ( Site 0323), Johannesburg, Gauteng
  - Albert Alberts Stem Cell Transplant Centre ( Site 0324), Pretoria, Gauteng
  - Wits Clinical Research ( Site 0321), Soweto, Gauteng
- South Korea (2):
  - Severance Hospital Yonsei University Health System ( Site 0221), Seoul
  - Samsung Medical Center ( Site 0222), Seoul
- Spain (3):
  - Hospital Universitari Vall d Hebron ( Site 0432), Barcelona
  - Hospital Infantil Universitario Nino Jesus ( Site 0433), Madrid
  - Hospital Universitario La Paz ( Site 0434), Madrid
- University College London Hospitals NHS Foundation Trust ( Site 0454), London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Castellino SM, Giulino-Roth L, Harker-Murray P, Kahn JM, Forlenza C, Cho S, Hoppe B, Parsons SK, Kelly KM; COG Hodgkin Lymphoma Committee. Children's Oncology Group's 2023 blueprint for research: Hodgkin lymphoma. Pediatr Blood Cancer. 2023 Sep;70 Suppl 6(Suppl 6):e30580. doi: 10.1002/pbc.30580. Epub 2023 Jul 28. PMID 37505794
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26281&tenant=MT_MSD_9011